CLINICAL TRIAL: NCT05286372
Title: An Intermediate Size, Expanded Access Protocol to Provide AMX0035, a Fixed Combination of Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO), for the Treatment of Adult Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: An Intermediate Size Expanded Access Protocol of AMX0035 for ALS
Status: Approved for marketing | Type: Expanded Access
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A35-006
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — sodium phenylbutyrate and taurursodiol

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: AMX0035 — Proprietary formulation of sodium phenylbutyrate and taurursodiol

SUMMARY:
The Expanded Access Program will provide access and assess the safety of AMX0035 for the treatment of people living with ALS.

DETAILED DESCRIPTION:
AMX0035 is a combination therapy designed to reduce neuronal death through blockade of key cellular death pathways originating in the endoplasmic reticulum (ER) and mitochondria. This Expanded Access Program is designed to provide expanded access to AMX0035 for the treatment of people living with ALS and assess safety in diverse populations/stages of ALS over 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age (inclusive);
* Diagnosis of ALS made by a physician experienced with the management of ALS;
* >36 months from symptom onset defined as first weakness
* Capable of providing informed consent;
* Capable of and willing to follow program procedures.
* Participants who have established care with a physician experienced in treating patients with ALS involved in the program and will maintain this clinical care throughout the duration of their time in the program.
* Women of childbearing potential (e.g., not post-menopausal for at least one year or surgically sterile) must agree to use adequate birth control for the duration of the program and 3 months after last dose of AMX0035;

  * Women must not be planning to become pregnant for the duration of the program and 3 months after last dose of study drug
* Men must agree to practice contraception for the duration of the program and for at least 3 months after last dose of program drug;

  * Men must not plan to father a child or provide sperm

Exclusion Criteria

* Currently enrolled in a therapeutic study involving the use of an investigational therapy;
* Dependence on invasive mechanical ventilation, defined as being unable to lay supine without it, unable to sleep without it, or continuous daytime use; presence of tracheostomy at Screening;

  * No current need for tracheostomy or PAV (defined as more than 22 hours daily of mechanical ventilation for more than one week (7 days) or based on the site investigator's judgment; no need anticipated for the next 12 weeks
* In the judgment of the Investigator, the participant's expected survival is less than 6 months
* History of known allergy to the following: PB, bile salts, excipient/constituents of the formulation;
* Abnormal liver function defined as AST and/or ALT >3 times the upper limit of the normal (obtained within 12 weeks from first dose);
* Renal insufficiency as defined by eGFR <60 mL/min/1.73m2 (obtained within 12 weeks from first dose);
* Pregnant women or women currently breastfeeding;
* Current severe biliary disease which may result in the investigator medical judgement in biliary obstruction including for example active cholecystitis, primary biliary cirrhosis, sclerosing cholangitis, gallbladder cancer, gallbladder polyps, gangrene of the gallbladder, abscess of the gallbladder;
* History of Class III/IV heart failure (per New York Heart Association - NYHA);
* Participant under severe salt restriction where the added salt intake due to treatment would put the participant at risk, in the Site Investigator clinical judgment;
* Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the participant to provide informed c consent, according to Site Investigator judgment;
* Clinically significant unstable medical condition (other than ALS) that would pose a risk to the participant if they were to participate in the program, according to Site Investigator judgment;
* Treatment, current or within 90 days from screening with any cell therapies or gene therapies;
* Implantation of Diaphragm Pacing System (DPS);
* Anything that, in the opinion of the Site Investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the program;
* Current or planned exposure to any prohibited medications listed in Section 6.8.1 of the protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (21):
- United States (20):
  - University of Southern California, Los Angeles, California
  - The Kaiser Permanente Medical Group, Oakland, California
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Holy Cross Health, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - The Sean M. Healey & AMG Center for ALS Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Neurology Associates, P.C. / Somnos Clinical Research, Lincoln, Nebraska
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Weinberg ALS Center, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - Providence St. Luke's Rehabilitation Medical Center, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
- Hispanic Alliance for Research & Translational Research, San Juan, Puerto Rico